CLINICAL TRIAL: NCT07171606
Title: A Phase II Study of SSGJ-706 Monotherapy and Combination Therapy in Advanced Non-Small Cell Lung Cancer（NSCLC） Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSGJ-706-201
Record Dates: First submitted 2025-09-01; First posted 2025-09-12 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-08

CONDITIONS: First-line Advanced NSCLC Patients
MeSH Terms: interventions — Pemetrexed; Carboplatin; CP protocol; Immune Checkpoint Inhibitors; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- dose level 1 of SSGJ-706 monotherapy (Experimental)
  Interventions: Drug: SSGJ-706
- dose level 2 of SSGJ-706 monotherapy (Experimental)
  Interventions: Drug: SSGJ-706
- dose level 1 of SSGJ-706 combined with chemotherapy (Experimental)
  Interventions: Drug: SSGJ-706; Drug: pemetrexed /carboplatin
- dose level 2 of SSGJ-706 combined with chemotherapy (Experimental)
  Interventions: Drug: SSGJ-706; Drug: Carboplatin/Paclitaxel
- PD-1/L1 combined with chemotherapy (Active Comparator)
  Interventions: Drug: PD-1 Inhibitor + Chemotherapy

INTERVENTIONS:
Drug: SSGJ-706 — PD-1/PD-L1 bispecific antibody
  Arms: dose level 1 of SSGJ-706 combined with chemotherapy; dose level 1 of SSGJ-706 monotherapy; dose level 2 of SSGJ-706 combined with chemotherapy; dose level 2 of SSGJ-706 monotherapy
Drug: pemetrexed /carboplatin — chemotherapy
  Arms: dose level 1 of SSGJ-706 combined with chemotherapy
Drug: Carboplatin/Paclitaxel — chemotherapy
  Arms: dose level 2 of SSGJ-706 combined with chemotherapy
Drug: PD-1 Inhibitor + Chemotherapy — control group
  Arms: PD-1/L1 combined with chemotherapy

SUMMARY:
This study includes two parts, part 1 is SSGJ-706 monotherapy therapy for advanced NSCLC and part 2 is SSGJ-706 combination therapy for advanced NSCLC

DETAILED DESCRIPTION:
This study is a study of SSGJ-706 monotherapy and combination therapy for advanced NSCLC Patients. This study includes two parts, part 1 is SSGJ-706 monotherapy therapy for advanced NSCLC and part 2 is SSGJ-706 combination therapy for advanced NSCLC. Each part will assess the efficacy and safety of the preset several dose levels of SSGJ-706 in advanced NSCLC Patients.

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or females over age 18
2. Histologically and/or cytologically documented local advanced or metastatic NSCLC .
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Expected survival >=3 months.
5. Signed informed consent form.

Exclusion Criteria:

1. Known uncontrolled or symptomatic central nervous system metastatic disease.
2. Adverse events (with exception of alopecia and fatigue) from any prior anticancer therapy of grade >1 (National Cancer Institute Common terminology Criteria [NCI CTCAE] v.5.0).
3. Inadequate organ or bone marrow function.
4. Pregnant or breast-feeding woman.
5. Known allergies, hypersensitivity, or intolerance to SSGJ-706

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 12 months
Incidence and severity of Adverse Events | 12 months

SECONDARY OUTCOMES:
DCR : Disease Control Rate | 12 months
PFS：Progression-Free Survival | 24 month
OS：Overall Survival | 24 month
The blood concentration of SSGJ-706 | Approximately 6 months
The incidence of Anti-drug antibody(ADA) and Neutralizing antibody(Nab) | Approximately 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of The Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No